CLINICAL TRIAL: NCT03171519
Title: Effects of Exercise and Acupuncture on Chronic Insomnia: a Randomized Control Trial
Brief Title: Effects of Exercise and Acupuncture on Chronic Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giselle Soares Passos, Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.998.334
Record Dates: First submitted 2017-05-18; First posted 2017-05-31 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Chronic Insomnia
Keywords: Physical activity; Disorders of onset and maintenance of sleep; non-pharmacological treatment; Acupuncture
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity | interventions — Exercise; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- Exercise + acupuncture (Experimental)
  Interventions: Behavioral: Exercise; Behavioral: Acupuncture

INTERVENTIONS:
Behavioral: Exercise — The EXERCISE group will participate in an aerobic exercise program for 12 weeks, performed in intensity relative to 50% of reserve heart rate, on a treadmill.
Behavioral: Acupuncture — The ACUPUNCTURE group will participate in an aerobic exercise program following the protocol of the EXERCISE group, plus acupuncture therapy once a week.
  Arms: Exercise + acupuncture

SUMMARY:
Introduction: Chronic insomnia is a sleep disorder, characterized by difficulty in initiating and/or maintaining sleep, presence of non-restorative sleep, frequent awakenings or difficulty returning to sleep after each awakening, with a frequency of 3 nights/week, for at least 3 months. Pharmacologic therapy is the most commonly method used for its treatment, however, pharmacotherapy is associated with side effects. Thus, non-pharmacological therapies have been suggested as an alternative. Objective: To verify the effects of exercise associated with acupuncture on chronic insomnia. METHODS: 40 patients with chronic insomnia will be randomly assigned into two groups: CONTROL (n = 20) and ACUPUNCTURE (n = 20). The volunteers of the CONTROL group will be submitted to 12 weeks of aerobic exercise, performed on a treadmill, with frequency of 3 times / week and duration of 50 minutes / day. ACUPUNCTURE volunteers will perform aerobic exercise, following the protocol of the CONTROL group, plus acupuncture therapy once a week. The sleep evaluation will be evaluated by polysomnography and questionnaires. Expected Results: A 12-week combined therapy could potentiate the previously described positive effects of exercise in the treatment of chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

* age 30-60 years;
* clinical diagnosis of chronic insomnia according to the DSM-V (performed by a physician specialized in Sleep Medicine);
* insomnia complaint at least 3 times a week for at least 3 months;
* be physically inactive (exercise less than 2 times a week).

Exclusion Criteria:

* evidence that insomnia is directly related to medical conditions or side effects os medications;
* obstructive sleep apnea syndrome;
* ECG abnormalities that prevent physical exercise or use of beta-blockers;
* uncontrolled clinical diseases (diabetes, hypertension, cardiovascular, neurological or renal diseases);
* use or history of abuse of alcohol or psychoactive substances;
* use of sleeping pills>2 times a week;
* shift workers.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline polysomnography to 12 weeks | baseline, week 12
  Polysomnographic recording included an electroencephalogram, an electrooculogram, an electromyogram, and an electrocardiogram. Measurements of air flow (oral and nasal), respiratory effort (thoracic and abdominal), body movement, and oxygen saturation were also taken. The measured variables included total sleep time, sleep efficiency (ratio between total sleep time and total recorded time multiplied by 100), sleep onset latency, wake after sleep onset, arousals, sleep stages (N1, N2 and N3 non-rapid eye movement [non-REM] sleep and REM sleep), latencies for each sleep stage. Two researchers who were blinded to the study design performed the staging and analysed the polysomnographic events using international criteria
Change from baseline anxiety to 12 weeks | baseline, week 12
  Prior sleep state anxiety will be assessed with the State-Trait Anxiety Inventory-STAI,25 the Portuguese version of which was validated by Gorenstein and Andrade.26 This scale encompasses 20 items and provides a one-dimensional measurement of anxiety. The volunteers were instructed to answer it 30 minutes before going to sleep at baseline and at the post-exercise evaluation.
Change from baseline mood to 12 weeks | 12 weeks
  The POMS questionnaire is an instrument to evaluate the acute profile of mood. It has 65 items and 6 domains: tension-anxiety, depression, anger-hostility, vigour-activity, fatigue, and confusion- bewilderment. The total mood disturbance score is derived by subtracting the vigour-activity score from the the sum of scores from the other subscales
Change from baseline sleep quality to 12 weeks | baseline, 12 weeks
  The PSQI assesses sleep quality over a 1-month period. The questionnaire consists of 19 self-rated questions and 5 questions that should be answered by bedmates or roommates. The latter questions are used only for clinical information. The 19 questions are categorized into 7 components, graded on a score that ranges from 0 to 3. The PSQI components are as follows: subjective sleep quality (C1), sleep latency (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disturbances (C5), use of sleeping medication (C6) and daytime dysfunction (C7). The sum of scores for these 7 components yields one global score, which ranges from 0 to 21, where the highest score indicates worst sleep quality. A global PSQI score greater than 5 indicates major difficulties in at least 2 components or moderate difficulties in more than 3 components.
Change from baseline quality of life to 12 weeks | baseline, week 12
  The SF-36 is a multidimensional questionnaire that covers eight components: physical functioning, role limitations due to physical health problems, role limitations due to emotional health problems, social functioning, vitality, general health perception, body pain, and mental health. All scores ranged from 0 to 100, with a higher score indicating better quality of life
Change from baseline insomnia to 12 weeks | baseline, week 12
  Insomnia Severity Index (ISI) was administrated at baseline and post treatment to assess insomnia-related complaints. It is a short and easy self-applied scale with 7 items scored from 0 to 4, with a total score varying from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia
Change from baseline sleep diary to 12 weeks | baseline, week 12
  The sleep diary was used to evaluate the subjective perceptions of sleep. Participants were instructed to complete the diary every morning after waking for 1 week. The parameters evaluated were sleep onset latency, wake after sleep onset, total time in bed, number of arousals, sleep quality, feeling rested in the morning, and sleep efficiency (calculated retrospectively by the researchers as the ratio of reported total sleep time and reported total time in bed multiplied by 100 [9]). These data were averaged for each volunteer for pre- and post-treatment assessment weeks.

SECONDARY OUTCOMES:
Change from baseline serum serotonin to 12 weeks | baseline, 12 weeks
  The blood sample will be collected at 8a.m. The serum serotonin dosage will be made by high performance liquid chromatography (HPLC)
Change from baseline cortisol to 12 weeks | baseline, 12 weeks
  The blood sample will be collected at 8a.m. The cortisol dosage will be made by chemiluminescence.
Change from baseline Effort eletrocardiogram test to 12 weeks | baseline, 12 weeks
  The test will be performed on a treadmill according to the protocol of Bruce.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Padre Thiago, Jatai, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided